

## Study protocol

Version 9; June 24th, 2022

# Comparison of McGrath Videolaryngoscopy and Direct Laryngoscopy for Rapid Sequence Intubation: an international, multicenter randomized trial

Kurt Ruetzler, MD<sup>1,2</sup>, , Yasin Tire, MD<sup>3</sup>, Gokhan Sertcakacilar, MD<sup>4</sup>, Elyad Ekrami, MD<sup>1</sup>, Edward Mascha, PhD<sup>1,5</sup>, and colleagues

- Department of OUTCOMES RESEARCH, Anesthesiology Institute, Cleveland Clinic, Cleveland, USA
- 2. Department of General Anesthesiology, Anesthesiology Institute, Cleveland Clinic, Cleveland, USA
- 3. The University of Health Science, Konya City Hospital, Konya Turkey
- 4. The University of Health Science, Bakırköy Dr. Sadi Konuk Education, and Research Hospital, Istanbul, Turkey
- 5. Department of Quantitative Health Sciences, Cleveland Clinic, Cleveland, USA

Address correspondence to: Kurt Ruetzler, M.D.; Department of OUTCOMES RESEARCH; Anesthesiology Institute; Cleveland Clinic; 9500 Euclid Avenue, P-77; Cleveland, Ohio, 44195; Telephone: (216)-445-9857, fax (216) 444-6135; E-mail: kr@or.org

On the World Wide Web: www.OR.org

### **BACKGROUND**

Securing the airway is a fundamental priority in the treatment of critically ill or injured patients. In the regular OR setting, direct laryngoscopy is the primary method for performing endotracheal intubation. But even in experienced hands, along with regular training and practice, successful endotracheal intubation sometimes requires additional tools to assist endotracheal intubation. Airway complications are rare but may lead to severe complications, such as brain damage and even death. Set aside the "cannot ventilate and cannot intubation" scenario, difficult intubation has been associated with significant patient morbidity. For example, repeated intubation attempts are associated with respiratory and hemodynamic complications, including hypoxemia, cardiac arrest, regurgitation, aspiration, and airway trauma — along with bradycardia and cardiac arrest in emergency settings 6.

Rapid Sequence Intubation (RSI) is indicated when patients are not fully conscious or are otherwise at increased risk of gastric regurgitation and aspiration.<sup>7</sup> The main objective of this technique is to minimize the time interval between loss of protective airway reflexes and tracheal intubation with a cuffed endotracheal tube. The period between induction of general anesthesia and securing the airway is most critical since aspiration of gastric content is then most likely.<sup>8</sup> However, rapid sequence induction is associated with, hemodynamic instability and oxygen desaturation.<sup>9-11</sup> It's therefore crucial to minimize the number of intubations attempts and the time to intubation, as both prolonged time to intubation and multiple intubation attempts significantly attribute to perioperative morbidity and mortality.

Videolaryngoscopes were introduced into clinical practice approximately two decades ago and have gained wide acceptance in the elective OR setting.<sup>12</sup> Videolaryngoscopes can facilitate endotracheal intubation by improving visualization of the larynx, thereby facilitating direct observation of the tracheal tube during passage through the vocal cords.<sup>13-17</sup> Consequently, videolaryngoscopy may decrease intubation difficulties and ultimately increase first-attempt and overall intubation success rate.<sup>13-17</sup> However,

available literature is heterogeneous in study design, patient characteristics, and intubation provider experience.

Several trials demonstrated that videolaryngoscopes improve vocal cord visualization, but not first-pass intubation success. <sup>18,19</sup> Interestingly, in a trial with ICU patients, videolaryngoscopy did not improve first-attempt intubation success and was associated with severe complications including death, cardiac arrest, cardiovascular collapse and hypoxemia. <sup>19</sup> In contrast, other trials reported improved glottis visualization, improved first-pass success <sup>16</sup> and no difference in rate of complications compared with direct laryngoscopy. <sup>20</sup> In a recent Cochrane review of more than seven thousand patients with and without difficult airways, videolaryngoscopy was associated with fewer complications (e.g., laryngeal or airway trauma, postoperative hoarseness, hypoxia), fewer failed intubations, and no increase in the time required for intubation. <sup>21</sup> The extent to which videolaryngoscopes might facilitate intubation in patients undergo RSI is unclear.

The McGrath (Medtronic, Minneapolis, MN) is an FDA-approved and commercially available videolaryngoscope that includes a Macintosh blade and a camera which provides an indirect view of the glottis. The McGrath has been tested in a variety of settings<sup>22-24</sup> and consistently provides better glottis visualization than direct laryngoscopy in patients with difficult airways.<sup>25,26</sup> However, its suitability in the context of RSI has yet to be formally evaluated, and whether results from previous trials apply to these patients remains unknown.

## **Objectives and Hypothesis**

Our goal is to compare conventional direct laryngoscopy using a Macintosh blade with the McGrath videolaryngoscope for rapid sequence endotracheal intubation. Specifically, we propose to test the *primary hypothesis* that videolaryngoscopy improves visualization of the vocal cords, defined using the modified Cormack and Lehane classification (primary outcome), versus direct laryngoscopy.

We will also test the <u>secondary hypotheses</u> that McGrath videolaryngoscopy decreases number of intubation attempts and the number of intubation failures. We hypothesize that the McGrath videolaryngoscopy reduces both, the number of intubation attempts and the number of intubation failures.

We will also assess the following exploratory outcomes:

- 1. Ease of intubation;
- 2. Glottis opening score (POGO) score;
- 3. Duration of intubation.

We will also assess the following safety outcomes:

- 1. Incidence of cut lips, airway injury, or dental injury;
- 2. Incidence of postoperative coughing;
- 3. Incidence or severity of postoperative sore throat;
- 4. Incidence or severity of postoperative hoarseness.

### **METHODS**

### Design

We propose a patient-blind multi-center randomized trial that will be coordinated by the Department of Outcomes Research at the Cleveland Clinic, Main Campus.

#### **Patients**

We will enroll up to 800 (including 25-50 pilot) consenting adults, with American Society of Anesthesiologists (ASA) physical status 1-3, who are scheduled for elective non-cardiac surgery requiring endotracheal intubation with rapid sequence induction for general anesthesia. Written informed consent will be obtained. Participating study centers will be:

- Cleveland Clinic, Main Campus, Cleveland OH
- Tabriz University of Medical Sciences, Tabriz, Iran
- · The University of Health Science, Konya City Hospital, Konya, Turkey
- The University of Health Science, Bakırköy Dr. Sadi Konuk Education, and Research Hospital, Istanbul, Turkey

# Inclusion criteria

- 1. Age between 18 and 99 years;
- 2. American Society of Anesthesiologists (ASA) physical status 1-3;
- 3. Elective surgery requiring oral endotracheal intubation for general anesthesia;
- 4. Any clinical indication for rapid sequence induction as determined by the attending anesthesiologist;
- 5. Anticipated extubation in the operating room.

# Exclusion criteria

- 1. Refusal of participation by attending anesthesiologist;
- 2. Indicated fiberoptic awake intubation

3. Body Mass index (BMI) > 45 kg/m<sup>2</sup>.

### **Protocol**

In the preoperative period, airway details for participating patients will be recorded by a research coordinator or anesthesia provider. Patients will be positioned supine and in a standardized ramped position on the OR table. Patients will be premedicated with midazolam, as clinically appropriate. All patients will be pre-oxygenated until the fraction of expired oxygen exceeds 80%.

Rapid sequence induction will be induced as preferred by the attending anesthesiologist, usually with a combination of lidocaine 1 mg/kg, propofol 2-5 mg/kg, fentanyl 1-3  $\mu$ g/kg, and succinylcholine 1.5 mg/kg or rocuronium 1.0 mg/kg. Complete muscle relaxation will be confirmed by absence of palpable twitches in response to supra-maximal train-of-four stimulation of the ulnar nerve at the wrist.

Patients will be randomized 1:1 before induction, stratified for primary anesthesia providers (*experienced* – specialist, attending *vs. unexperienced* – trainees) to:

- <u>Direct laryngoscopy</u> using an appropriately sized Macintosh blade (usually size 3 or 4);
- McGrath videolaryngoscope in an appropriate size (usually blade size 3 or 4).

Randomization will be based on computer-generated codes accessed from the Redcap system.

Intubations will be performed with a regular endotracheal tube of adequate diameter, usually 7.0 mm to 8.0 mm. Endotracheal tubes will be equipped with a hockey-stick-shaped stylette, which will be prepared by the anesthesiologist in advance. The McGrath or the Macintosh blade will be introduced into oral cavity according to manufacturer recommendations and clinical practice. Minor airway manipulation procedures including BURP or Sellick maneuvers will be allowed to improve

visualization of the vocal cords. If initial intubation attempts fail, the endotracheal tube will be removed. Minor adjustments of patient's position and/or tube stylette will be used as clinically appropriate. Up to two intubation attempts will be made as necessary. Further airway management will follow clinical assessment of the anesthesiologist. The anesthesiologist will be permitted to terminate study participation and switch to an alternative method.

Once intubation is achieved, the endotracheal tube will be connected to the anesthesia circuit, and the endotracheal cuff pressure will be measured placed between 25 and 30 cm  $H_2O$ .

Mechanical ventilation with  $O_2$  and air will be adjusted to maintain end-tidal PCO<sub>2</sub> between 32 and 35 mmHg as clinically necessary. Maintenance of general anesthesia will be provided, as clinically indicated.

At the end of the surgical procedure, patients will be extubated and transferred to the post anesthesia care unit (PACU). Patients will then be assessed for postoperative complications 2 hours following extubation, or at PACU discharge.

## Measurements

Demographic and morphometric characteristics will be collected from electronic medical records.

- 1. Age
- 2. Sex
- 3. Race
- 4. BMI
- 5. ASA status
- 6. Airway examination
  - a. History of obstructive sleep apnea (yes/no)
  - b. History of snoring (yes/no)

- c. History of CPAP (yes/no)
- d. History of difficult airway (yes/no)
- e. Mobility of cervical spine (0, 15, 30, and 45 degrees)
- f. Mouth opening (cm)
- g. Inter-incisor gap (cm)
- h. Mandibular protrusion test (Class A, B, C)
- i. Thyro-mental distance (cm)
- j. Thyro-mental height (cm)
- k. Sterno-mental distance (cm)
- I. Neck circumference (cm)
- m. Upper lip bite test (Class I, II, III)
- n. Mallampati score (1/2/3/4)
- o. Teeth status (Edentulous, missing frontal teeth or full dentition)

# Outcomes

# Primary outcome:

Best glottis visualization, defined as visualization according to the modified Cormack and Lehane classification<sup>27</sup>

| | 1 | 2 Partial view of the glottis or arytenoids | | 3<br>Only epiglottis<br>visible | 4<br>Neither glottis nor<br>epiglottis visible |
|---|---|---|---|---|---|
| Original Cormack<br>and Lehane system<br>View at<br>laryngoscopy | Full view of the glottis | | | | |
| | | 8 | | | |
| Modified system | 1<br>As for original<br>Cormack and<br>Lehane above | 2a<br>Partial view of the<br>glottis | 2b Arytenoids or posterior part of the vocal cords only just visible | 3 As for original Cormack and Lehane above | 4<br>As for original<br>Cormack and<br>Lehane above |

## Secondary Outcomes:

- Intubation attempts, defined as introducing the endotracheal tube into oral cavity to perform endotracheal intubation (1, 2, 3, etc.)
- · Intubation failure, defined as
  - Failure to intubate within 3 intubation attempts
  - Need to switch intubators or intubation device
  - Need to stop study per anesthesiologist's discretion

# Exploratory outcomes:

- Portion of glottis opening score (POGO) score, defined as estimation of the glottis, which is visible during laryngoscopy (0, 25, 50, 75, 100%)<sup>28,29</sup>
- Time to intubation, defined as the time between the laryngoscope introduced into oral cavity and cuff inflation (RSI definition) and to the first appearance of endtidal CO<sub>2</sub>.
- Ease of intubation, defined as subjective evaluation of the anesthesiologist after finishing the intubation procedure: (1) very easy; (2) easy; (3) moderate;
   (4) difficult; and, (5) impossible.<sup>30,31</sup>

# Safety outcomes:

- Any apparent airway or dental injury including bleeding, airway trauma, dental fracture, aspiration, or bronchospasm.
- Incidence and severity of postoperative cough, assessed 2 hours after extubation in the PACU, and defined as continuous throat pain and rated as mild (less than a common cold), moderate (similar to a common cold), or severe (more than a common cold).<sup>30,31</sup>

- Incidence and severity of postoperative sore throat, assessed after 2 hours of
  extubation in the PACU, defined as an acoustic quality that was different from the
  previous voice quality of the patients and rated as mild (less than a common
  cold), moderate (similar to a common cold), or severe (more than a common
  cold).<sup>30,31</sup>
- Incidence and severity of postoperative hoarseness, assessed after 2 hours of extubation in the PACU, and rated as noticed by the patient only, apparent to an observer, or aphonia.<sup>30,31</sup>

### Data analysis:

### Statistical Analysis

We will assess the balance of two randomized groups (McGrath videolaryngoscopy vs. direct laryngoscopy) on **baseline and demographic characteristics** using the absolute standardized difference (ASD), defined as the absolute difference in means, mean ranks, or proportions divided by the pooled standard deviation. Any characteristics with ASD > maximum of 0.10 and  $1.96\sqrt{(n_1n_2)x(n_1+n_2)}$  will be considered imbalanced and will be adjusted for in the primary and secondary analyses.

All primary and secondary analyses will be completed using the modified intent-to-treat principle, thus including all randomized patients in whom intubation was attempted in the analyses. We will conservatively assign all missing outcome values as the highest possible score in the control group (direct laryngoscopy) and the lowest possible score in the treatment group (McGrath videolaryngoscopy) for all primary and secondary analyses.

### Primary outcome:

Wilcoxon-Mann-Whitney test will be used to formally compare categorical outcome of glottis visualization (Cormack and Lehane classification) at the 5% significance level

Formatted: Font: Bold

between the two study groups; this test accounts for the ordinal nature of the outcome. If adjustment for imbalanced baseline covariates is required, we will attempt a proportion odds logistic regression model to compare randomized groups, reporting an odds ratio indicating the estimated odds of being better using videolaryngoscopy versus direct.

**Commented [WP1]:** See <u>here</u> for details on implementation and diagnostics.

If the proportional odds assumption does not hold after testing and also visualizing with further modeling, the outcome will be assessed using either an adjacent logit analysis or by combining categories and using chi-square test or binary logistic regression, as appropriate. The distribution of patients in each glottis visualization class will be reported for each randomized group.

Commented [WP2]: In `vgam` R package, the `acat()` function.

Commented [WP3R2]: Response MUST be an ordered factor. Returns an object of class vglmff to be used by vgam/vglm

# Secondary outcomes:

Randomized groups will be compared on the secondary outcome of Intubation failure (yes/no) via chi-square test and the associations reported using relative risk [97.5% confidence interval (CI)]. Randomized groups will be compared on the count of number of intubation attempts using either Wilcoxon-Mann-Whitney test or negative binomial regression, as appropriate. A Bonferroni correction will be applied and a significance criterion of 0.05/2=0.025 to control the overall Type I error at 5% level for two secondary hypotheses.

The exploratory and safety outcomes will be reported by study groups without formal statistical testing of the difference.

Formatted: Highlight

**Interim analyses** to assess efficacy and futility will be conducted at each 25% of the maximum planned enrollment. We will use a gamma spending function with gamma parameter= -4 for efficacy and -1 for futility.

Sample size considerations. Sample size is based on the primary outcome of glottis visualization (Cormack and Lehane classification) and the Wilcoxon-Mann-Whitney test. From the literature we assume a distribution of scores for the Direct Laryngoscopy group such that the proportion of patients in categories 1, 2a, 2b, 3 and 4 are 0.50, 0.30, 0.15, 0.04, 0.01, and that for the videolaryngoscopy the proportions are improved to 0.65, 0.25, 0.07, 0.02, 0.01. We would thus need a total of 384 patients to detect this difference or larger with 90% power at the 0.05 significance level. Incorporating a maximum of 3 interim analyses and a final analysis with the above-detailed spending functions will require a maximum of N=438 patients. Simulations indicate that if the specified difference is a good estimate of the true effect, the expected sample size is about 78% of the maximum sample size, or N=342. In such a case, the study will have a very good chance of crossing an efficacy boundary at interim looks 2 or 3.

Because our estimates of laryngeal view are uncertain, we plan to enroll a maximum of 800 patients in case the treatment effect is somewhat less than anticipated.

**Pilot patients:** We will enroll 5-10 pilot patients prior to the start of the study at each study center to familiarize the study team with the protocol and identify any systematic issues that might result in protocol modifications. Pilot patients will be randomized either to McGrath videolaryngoscopy or direct laryngoscopy group in the same manner as it is planned for the study. Pilot patients will not be included in the statistical analysis.

# **Funding:**

This study is an investigator-initiated study.

Formatted: Font color: Red

Formatted: Font color: Red

Formatted: Font color: Light Blue

Formatted: Font color: Red

### **REFERENCES**

- 1. Wang HE, Seitz SR, Hostler D, Yealy DM: Defining the learning curve for paramedic student endotracheal intubation. Prehosp Emerg Care 2005; 9: 156-62
- 2. Garza AG, Gratton MC, Coontz D, Noble E, Ma OJ: Effect of paramedic experience on orotracheal intubation success rates. J Emerg Med 2003; 25: 251-6
- 3. Deakin CD, King P, Thompson F: Prehospital advanced airway management by ambulance technicians and paramedics: is clinical practice sufficient to maintain skills? Emerg Med J 2009; 26: 888-91
- 4. Cook TM, MacDougall-Davis SR: Complications and failure of airway management. Br J Anaesth 2012; 109 Suppl 1: i68-i85
- 5. Hasegawa K, Shigemitsu K, Hagiwara Y, Chiba T, Watase H, Brown CA, 3rd, Brown DF: Association between repeated intubation attempts and adverse events in emergency departments: an analysis of a multicenter prospective observational study. Ann Emerg Med 2012; 60: 749-54.e2
- 6. Mort TC: Emergency tracheal intubation: complications associated with repeated laryngoscopic attempts. Anesth Analg 2004; 99: 607-13, table of contents
- 7. El-Orbany M, Connolly LA: Rapid sequence induction and intubation: current controversy. Anesth Analg 2010; 110: 1318-25
- 8. Olsson GL, Hallen B, Hambraeus-Jonzon K: Aspiration during anaesthesia: a computer-aided study of 185,358 anaesthetics. Acta Anaesthesiol Scand 1986; 30: 84-92
- 9. Gebremedhn EG, Mesele D, Aemero D, Alemu E: The incidence of oxygen desaturation during rapid sequence induction and intubation. World J Emerg Med 2014; 5: 279-85
- 10. Higgs A, McGrath BA, Goddard C, Rangasami J, Suntharalingam G, Gale R, Cook TM: Guidelines for the management of tracheal intubation in critically ill adults. Br J Anaesth 2018; 120: 323-52
- 11. Ahmed A, Azim A: Difficult tracheal intubation in critically ill. J Intensive Care 2018; 6: 49

- 12. Weiss MS, U.; Gerber, AC.: Video-Intubating Laryngoscopy A New concept four Routine and Difficult Tracheal Intubation Management. Anesthesiology 1998; Suppl. 3A, SEE9
- 13. Aziz MF, Abrons RO, Cattano D, Bayman EO, Swanson DE, Hagberg CA, Todd MM, Brambrink AM: First-Attempt Intubation Success of Video Laryngoscopy in Patients with Anticipated Difficult Direct Laryngoscopy: A Multicenter Randomized Controlled Trial Comparing the C-MAC D-Blade Versus the GlideScope in a Mixed Provider and Diverse Patient Population. Anesth Analg 2015
- 14. Piepho T, Fortmueller K, Heid FM, Schmidtmann I, Werner C, Noppens RR: Performance of the C-MAC video laryngoscope in patients after a limited glottic view using Macintosh laryngoscopy. Anaesthesia 2011; 66: 1101-5
- 15. Sakles JC, Mosier J, Chiu S, Cosentino M, Kalin L: A comparison of the C-MAC video laryngoscope to the Macintosh direct laryngoscope for intubation in the emergency department. Ann Emerg Med 2012; 60: 739-48
- 16. Aziz MF, Dillman D, Fu R, Brambrink AM: Comparative Effectiveness of the C-MAC Video Laryngoscope versus Direct Laryngoscopy in the Setting of the Predicted Difficult Airway. Anesthesiology 2012; 116: 629-36
- 17. Jungbauer A, Schumann M, Brunkhorst V, Borgers A, Groeben H: Expected difficult tracheal intubation: a prospective comparison of direct laryngoscopy and video laryngoscopy in 200 patients. Br J Anaesth 2009; 102: 546-50
- 18. Sulser S, Ubmann D, Schlaepfer M, Brueesch M, Goliasch G, Seifert B, Spahn DR, Ruetzler K: C-MAC videolaryngoscope compared with direct laryngoscopy for rapid sequence intubation in an emergency department: A randomised clinical trial. Eur J Anaesthesiol 2016; 33: 943-8
- 19. Lascarrou JB, Boisrame-Helms J, Bailly A, Le Thuaut A, Kamel T, Mercier E, Ricard JD, Lemiale V, Colin G, Mira JP, Meziani F, Messika J, Dequin PF, Boulain T, Azoulay E, Champigneulle B, Reignier J: Video laryngoscopy vs direct laryngoscopy on successful first-pass orotracheal intubation among icu patients: A randomized clinical trial. Jama 2017; 317: 483-93
- 20. Taylor AM, Peck M, Launcelott S, Hung OR, Law JA, MacQuarrie K, McKeen D, George RB, Ngan J: The McGrath(R) Series 5 videolaryngoscope vs the

Macintosh laryngoscope: a randomised, controlled trial in patients with a simulated difficult airway. Anaesthesia 2013; 68: 142-7

- 21. Lewis SR, Butler AR, Parker J, Cook TM, Smith AF: Videolaryngoscopy versus direct laryngoscopy for adult patients requiring tracheal intubation. Cochrane Database Syst Rev 2016; 11: Cd011136
- 22. Kwak HJ, Lee SY, Lee SY, Cho SH, Kim HS, Kim JY: McGrath Video Laryngoscopy Facilitates Routine Nasotracheal Intubation in Patients Undergoing Oral and Maxillofacial Surgery: A Comparison With Macintosh Laryngoscopy. J Oral Maxillofac Surg 2016; 74: 256-61
- 23. Hyuga S, Sekiguchi T, Ishida T, Yamamoto K, Sugiyama Y, Kawamata M: Successful tracheal intubation with the McGrath((R)) MAC video laryngoscope after failure with the Pentax-AWS in a patient with cervical spine immobilization. Can J Anaesth 2012; 59: 1154-5
- 24. Foulds LT, McGuire BE, Shippey BJ: A randomised cross-over trial comparing the McGrath((R)) Series 5 videolaryngoscope with the Macintosh laryngoscope in patients with cervical spine immobilisation. Anaesthesia 2016; 71: 437-42
- 25. Noppens RR, Mobus S, Heid F, Schmidtmann I, Werner C, Piepho T: Evaluation of the McGrath Series 5 videolaryngoscope after failed direct laryngoscopy. Anaesthesia 2010; 65: 716-20
- 26. Shippey B, Ray D, McKeown D: Use of the McGrath videolaryngoscope in the management of difficult and failed tracheal intubation. Br J Anaesth 2008; 100: 116-
- 27. Yentis SM, Lee DJ: Evaluation of an improved scoring system for the grading of direct laryngoscopy. Anaesthesia 1998; 53: 1041-4
- 28. Biro P, Ruetzler K: The reflective intubation manoeuvre increases success rate in moderately difficult direct laryngoscopy: A prospective case-control study. Eur J Anaesthesiol 2015; 32: 406-10
- 29. Cormack RS, Lehane JR, Adams AP, Carli F: Laryngoscopy grades and percentage glottic opening. Anaesthesia 2000; 55: 184-

- 30. Ruetzler K, Grubhofer G, Schmid W, Papp D, Nabecker S, Hutschala D, Lang G, Hager H: Randomized clinical trial comparing double-lumen tube and EZ-Blocker for single-lung ventilation. Br J Anaesth 2011; 106: 896-902
- 31. Ruetzler K, Guzzella SE, Tscholl DW, Restin T, Cribari M, Turan A, You J, Sessler DI, Seifert B, Gaszynski T, Ganter MT, Spahn DR: Blind intubation through self-pressurized, disposable supraglottic airway laryngeal intubation masks: An international, multicenter, prospective cohort study. Anesthesiology 2017; 127: 307-16